CLINICAL TRIAL: NCT01918228
Title: Effect of an Educational Based Intervention on Danish Workers With Low Back Pain. A Randomized Controlled Single Blinded Study.
Brief Title: Effect of Reassuring Information on Danish Workers Who Experience Low Back Pain in the Following Year.
Acronym: VRRPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: National Research Centre for the Working Environment, Denmark (Other Government); University of Huddersfield (Other); University of Bergen (Other)
Responsible Party: Principal Investigator, Pernille Frederiksen, PhD Student, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: VRRPhDPF; PF2013 (Registry Identifier: Pernille Frederiksen)
Record Dates: First submitted 2013-04-25; First posted 2013-08-07 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Non-specific Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Talks on scientific status on back pain with the purpose of reducing LBP-related insecurity/fear, reducing the focus on the pain and providing participants with alternative explanation to their LBP. They were also provided with a folder (general stretching exercises) and had telephone access to health professional if they had questions about LBP during the follow-up year.
  Interventions: Behavioral: Talks about what science says about LBP
- Control group (No Intervention): No intervention will be provided by the study team.

INTERVENTIONS:
Behavioral: Talks about what science says about LBP — Two talks, a folder with general stretching exercises and possibility to contact health professional by telephone
  Arms: Intervention group

SUMMARY:
RCT study of the effect of an educational-based intervention on low back pain-related outcomes concerning beliefs and behaviour.

DETAILED DESCRIPTION:
Previous studies have strongly implied that information is a valuable means for people suffering from LBP in terms of coping appropriately. Most studies have tested the effect of information as part of a multimodal intervention.

Four Nordic studies testing the effect of 'reassuring information' based on the 'Functional Disturbance'-model (proposed by Indahl et al. 1999 - also called the 'non-injury'-model) have all been effective at positively altering the functional level and/or days of sickness absence - when provided in combination with other elements to people with subacute/chronic back pain. The present study set out to test the effect of this kind of resassuring information alone.

Between November 2012 and September 2013, we included app. 500 municipal workers perfoming either manual work, administrative work or a combination of the two. Participants worked in 5 different municipal workplaces. These workplaces were characterized by being devided into 'natural working unit', which had no or very little daily contact. All 5 workplaces participated with at least 2 units. Thus 11 units contributed to the data. Baseline assessment took place during right upon recruitment prior to randomization.

We cluster-randomized the 11 units into an intervention and a control group using a simple stepwise randomization-metod.

The intervention group received two 45-minute lectures at the workplace with an interval of 2 weeks. The lectures were coherent allthough different. They consisted of information on the scientific knowledge on the etiology of LBP, basic anatomy, common myths about LBP, a theory of non-specific LBP being caused by muscular functional disturbances (Indahl 1999), pain physiology, and scientific knowledge on seemingly appropriate coping strategies to prevent a prolonged course. Emphasis was made to reduce pain-related fear of movement and catastrophizing thoughts and beliefs. Instead, activity during pain episodes was promoted as well as a natural use of the back despite pain. A non-directive approach was used (non-imperativ wording and absence of giving advice). The purpose was to provide information but let the participant make their own conclusions on how and if to use the information in present/future coping with pain.

In addition to the lecture, the intervention group participants were provided with a leaflet showing various relevenat stretching exercises (back and related muscles) and they were offered the option to make a call to the primary investigator in case any questions would arise subsequently.

The control group was untreated by us. Both groups had access to all 'usual' help (workplace, general practitioner etc).

Upon completion of the lectures, twelve monthly assessments were conducted using Text Messaging (SMS). During each assessment, participants answered questions on no. of LBP days, no. of LBP-related cutdown days, no. of LBP-related sick days, no. of LBP-related healthcare visits, overall workability, bothersomeness last week, restricted activity last week, and use of pain medicine or degree of sadness/depression.

In addition, a separate assessment was performed at app. 5.5 monts to obtain responses on back beliefs.

The data collection was completed in 2014. Analysis are nearly finished. The sicentific paper on the study is anticipated to take place in the beginning of 2016.

ELIGIBILITY:
Inclusion Criteria:

-employed at one of the participating municipal workplaces

Exclusion Criteria:

* pregnancy within the first 6 months of the study
* physical or mental disease that has significant impact on the individual in terms of pain (eg. Rheumathoid disease, clinical depression)
* present cancer disease (risk of metastasis)
* planned stop at the workplace within the first 6 months of the study

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Functional Level | 12 months
  item 2 & 4 in the COMI (Deyo et al. 1998) cathegoric variable/numeric variable
Sickness absence (analysed as work participation) | 12 months
  item 5 in the COMI (Deyo et al. 1998)

SECONDARY OUTCOMES:
No. of monthly healthcare visits | 12 months
  Number of monthly visits to any kind of healthcare provider
Back beliefs | 5.5 months
  item 10 & 12-14 from the Back Beliefs Questionnaire

OTHER OUTCOMES:
Overall Workability | 12 months
  single item from the Workability Index (WAI) numeric continuant variable,
Bothersomeness last week | 12 months
  item 2 from the COMI (Deyo et al. 1998)
Restricted activity last week | 12 months
  item 3 from the COMI (Deyo et al. 1998)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Bendix, Professor, Study Chair — Copenhagen Center for Back Research
Locations (1):
- Copenhagen Center for Back Research, Glostrup Municipality, Denmark